CLINICAL TRIAL: NCT02205125
Title: Prospective Characterization of the Mucosal Defect After Cold Snare Polypectomy
Brief Title: Cold Polypectomy Site Study
Status: Completed | Type: Observational
Sponsor: Professor Michael Bourke (Other)
Responsible Party: Sponsor-Investigator, Professor Michael Bourke, Director of Endoscopy, Westmead Hospital, Sydney, Australia, Western Sydney Local Health District
Organization: Western Sydney Local Health District (Other)
Other Study IDs: HREC2013/8/6.6(3797)
Record Dates: First submitted 2014-07-26; First posted 2014-07-31 (Estimated); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Colonic Polyps
Keywords: polyp; colon; polypectomy; snare
MeSH Terms: conditions — Colonic Polyps; Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — All polypectomy specimens were submitted for histopathological assessment as per clinical practice. The biopsy samples from the irregular areas were also submitted in the same fashion. All specimens are stored as per current clinical practice.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Removal of polyps at colonoscopy reduces colon cancer. Snare polypectomy is the conventional method for removal however the snared area after removal can occasionally appear uneven raising the possibility that complete removal has not occurred. The significance of this irregularity has not be studied. This study aims to separately sample the irregular area and determine the constituents while recording how frequently this occurs during routine colonoscopy and polypectomy. We hypothesize that the irregular areas are submucosal tissue and do not represent polyp tissue left behind.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing colonoscopy with at least one polyp identified where polypectomy is planned.

Exclusion Criteria:

* Age < 18 years
* Patients where polypectomy is not planned to be undertaken (patients scheduled for diagnostic colonoscopy only).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing colonoscopy at a tertiary endoscopy unit.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2013-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Frequency and constituents of stalk projections in cold snare polypectomy sites | 14 days
  Biopsy of post cold snare polypectomy stalk to determine constituents of stalk. This was reviewed 14 days following the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bourke, MBBS, FRACP, Principal Investigator — WSLHD
Locations (1):
- Westmead Hospital Endoscopy Unit, Sydney, New South Wales, Australia